CLINICAL TRIAL: NCT04217317
Title: Pilot Study of CPI-613, in Combination With Bendamustine, in Patients With Relapsed or Refractory T-Cell Non-Hodgkin Lymphoma
Brief Title: CPI-613 in Combination With Bendamustine in Patients With Relapsed/Refractory T-Cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00062873; WFBCCC 28419 (Other: IRB - Wake Forest University Health Science); P30CA012197 (NIH)
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Relapsed T-Cell Lymphoma; Refractory T-Cell Lymphoma; Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell; Lymphoma, Non-Hodgkin | interventions — devimistat; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-613 in Combination with Bendamustine (Experimental): CPI-613 at 2500 mg/m2 is infused intravenously (IV) via a central catheter over 2 hrs on Days 1and 2. Bendamustine at 90 mg/m2 is infused IV over 10 minutes on Days 1 and 2 of each treatment cycle, given immediately after CPI-613 administration.
  Interventions: Drug: CPI 613; Drug: Bendamustine

INTERVENTIONS:
Drug: CPI 613 — CPI-613 is to be given as 2-hr IV infusion via a central venous catheter. The starting dose of CPI-613 will be 2500 mg/m2 which was determined to be the MTD in the previous phase I clinical trial.
  Other Names: devimistat
Drug: Bendamustine — Bendamustine at 90 mg/m2 is infused by IV over 10 minutes on Days 1 and 2 of each treatment cycle. Bendamustine is given immediately after CPI-613 administration.
  Other Names: Bendeka; Treanda; Bendamustine Hydrochloride

SUMMARY:
The purpose of this study is to determine if it is possible to give CPI-613 with the drug Bendamustine for 2 days every 28 days without causing severe side effects. In addition, this study will also test the safety of CPI-613 when given in combination with Bendamustine.

DETAILED DESCRIPTION:
Primary Objectives: A pilot Study to evaluate the feasibility, safety and tolerability of a two day course per cycle of Bendamustine plus CPI-613 in patients with relapsed and refractory T cell non-hodgkin lymphoma.

Exploratory Objectives

To evaluate:

* Overall response rate (ORR) and disease control rate (DCR) derived from the Lugano classification.
* Duration of response (DOR) derived from the Lugano classification.
* Progression-Free-Survival (PFS) derived from Lugano classification.
* Overall Survival (OS).
* Single cell transcriptomics from PMBCs pre- and post-treatment; for correlative analyses of blood PBMC (and possibly excess pre-treatment tumor biopsy) cell population diversity and functional states to reveal potential mechanisms of drug treatment with regard to patient response status.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria before enrollment:
* Histologically or cytologically confirmed PTCL (all subtypes) or CTCL (mycosis fungoides/Sezary syndrome) as defined by 2016 World Health Organization (WHO) classification.

For patients with PTCL:

* Patients must have relapsed/refractory disease to one or more systemic therapies.
* Patients with CD30-positive lymphoma must have received, be ineligible for, or intolerant to brentuximab vedotin.
* Patients with limited prior exposure to Bendamustine (less than 2 full cycles or ≤ 480 mg/m2) may be included, based on PI discretion.
* Patients must have measurable disease (e.g., a tumor mass >1 cm or evidence of bone marrow involvement).

For patients with CTCL, Stage IB-IVB mycosis fungoides or Sezary syndrome are eligible

* Patients must have relapsed/refractory disease to at least one previous systemic therapy. Psoralen plus ultraviolet light therapy (PUVA) is not considered to be a systemic therapy.
* Male and female patients 18 years of age and older
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Expected survival greater than 3 months.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists.
* At least 2 weeks must have elapsed from prior chemotherapy drugs (other than steroids) or radiation
* At least 6 weeks must have elapsed from prior autologous stem cell transplant and 12 weeks must have elapsed from prior allogeneic stem cell transplant.
* Laboratory values ≤2 weeks must be: Adequate hematological function (absolute neutrophil count [ANC] ≥1,500/mm3, platelets ≥100,000/mm3). In subjects with known bone marrow involvement, ANC must be ≥ 1000/mm3 and platelets ≥75,000/mm3; Adequate hepatic function (aspartate aminotransferase [AST/SGOT] less than or equal to 3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] less than or equal to 3x UNL (≤5x UNL if liver metastases present), bilirubin less than or equal to 1.5x UNL); Adequate renal function (serum creatinine less than or equal to 1.5 mg/dL or 133 µmol/L).
* No evidence of current infection.
* Mentally competent, ability to understand and willingness to sign the informed consent form.

Exclusion Criteria:

* Patients with the following characteristics are excluded:
* Known cerebral metastases, central nervous system (CNS) or epidural tumor.
* History of prior malignancy and considered to be at greater than 30% risk of relapse
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of treatment with study drugs (steroids are allowed)
* Patients with a history of allogeneic transplant must not have ≥ grade 3 graft-versus-host disease (GVHD) or any clinically significant GVHD requiring systemic immunosuppression.
* Serious medical illness that would potentially increase patients' risk for toxicity.
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown).
* Lactating females.
* Fertile men unwilling to practice contraceptive methods during the study period.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
* Unwilling or unable to follow protocol requirements.
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction or symptomatic congestive heart failure.
* Evidence of current infection..
* Patients with known HIV infection, hepatitis B, or hepatitis C with positive viral load.
* Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2024-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakhee Vaidya, M.B.B.S., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CPI-613 in Combination With Bendamustine
Started | 6
Completed | 1
Not Completed | 5
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants To Successfully Complete Therapy Regimen
Description: Number of patients successfully able to complete 80% (at least 5 of 6 planned cycles) of their therapy regimens.
Time Frame: up to 6 cycles, up to 24 weeks after first dose
Measure: Count of Participants; unit: Participants
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the proportion of patients who achieve a best overall response complete response or partial response during or following study treatment.
  Response derived from the Lugano classification for PTCL patients and Global Response Score for CTCL (MF/SS) patients. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: The Lugano classification.
Time Frame: Patients are monitored for best overall response during and after study treatment. Follow-up for response ranged from 2 to 6 months after start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: Disease Control Rate
Description: Disease control rate defined as the proportion of patients who achieve a best overall response of complete response, partial response, or stable disease (SD). Best overall response of stable disease must have met the response stable disease criteria at least once ≥12 weeks after start of study treatment. Response derived from the Lugano classification for PTCL patients and Global Response Score for CTCL (MF/SS) patients
Time Frame: Patients are monitored for response during and after study treatment. Follow-up for response ranged from 2 to 6 months after start of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 6
Participants | 3

4. Secondary Outcome: Duration of Response
Description: Duration of Response will be defined for responders (patients with a best overall response of complete response or partial response). It is the time from the date of the first documented complete response or partial response until the date of the first date of progressive disease, or death due to any cause, whichever occurs first. If a patient has not progressed or died by the analysis cutoff date, duration of response will be censored at the time of the last adequate tumor assessment on or before the cutoff date.
  Response derived from the Lugano classification for PTCL patients and Global Response Score for CTCL (MF/SS) patients.
Time Frame: as for outcome 3
Population: patients who had a complete or partial response during the study.
Measure: Median (Full Range); unit: months
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 1
months | 2.3 [2.3 to 2.3]

5. Secondary Outcome: Progression Free Survival
Description: Progression free survival defined as the time from the start of study treatment until the first date of progressive disease, or death due to any cause, whichever occurs first. If a patient has not progressed or died by the analysis cutoff date, progression free survival will be censored at the time of the last adequate tumor assessment on or before the cutoff date.
  Response derived from the Lugano classification for PTCL patients and Global Response Score for CTCL (MF/SS) patients
Time Frame: Patients are monitored for progression during and after study treatment. Follow-up for response ranged from 2 to 6 months after start of treatment.
Measure: Median (Full Range); unit: months
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 6
months | 2.7 [2.1 to 6.1]

6. Secondary Outcome: Overall Survival
Description: Overall survival is measured from the start of study treatment until death due to any cause. If a patient is not known to have died at the date of the analysis cut-off, overall survival will be censored at the last date that: Patient is documented to be alive. At the time of single cell sequencing.
Time Frame: Maximum observed follow-up of 3 years 9 months
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | CPI-613 in Combination With Bendamustine
Number analyzed (Participants) | 6
months | 7.5 [6.5 to 17.1]

ADVERSE EVENTS:
Time Frame: Adverse events are monitored from the start of treatment until 30 days after last treatment dose. Average of 7.8 months with range of 16.6 months. The timeframe for all cause mortality is longer and has a maximum observed follow-up of 3 years 9 months.
Arm/Group | CPI-613 in Combination With Bendamustine
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPI-613 in Combination With Bendamustine (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations - Other: Catheter related infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPI-613 in Combination With Bendamustine (N=6)
Anemia (Blood and lymphatic system disorders) | 4 (9)
Cardiac disorders - Other: BASELINE MURMUR (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 4 (4)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Infections and infestations - Other: FUNGAL POSITIVE SPUTUM (Infections and infestations) | 1 (1)
Infections and infestations - Other: INCREASED MONOCYTES (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (5)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 5 (11)
Neutrophil count decreased (Investigations) | 3 (7)
Platelet count decreased (Investigations) | 3 (10)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (7)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (10)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (7)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (5)
Skin and subcutaneous tissue disorders - Other: Bumps on head and face (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other: NEW SKIN LESIONS (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT04217317/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04217317/ICF_000.pdf